CLINICAL TRIAL: NCT04916236
Title: Phase I/Ib Study With the Combination of RMC-4630 (SHP2 Inhibitor) and LY3214996 (ERK Inhibitor) in Metastatic KRAS Mutant CRC, PDAC and NSCLC
Brief Title: Combination Therapy of RMC-4630 and LY3214996 in Metastatic KRAS Mutant Cancers
Acronym: SHERPA
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to a lack of safety and efficacy.
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Lustgarten Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M20SHP
Record Dates: First submitted 2021-05-06; First posted 2021-06-07 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Pancreatic Cancer; Colorectal Cancer; Non-small Cell Lung Cancer; KRAS Mutation-Related Tumors
Keywords: SHP2; ERK; Combination therapy; KRAS mutation-related tumors
MeSH Terms: conditions — Pancreatic Neoplasms; Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — LY3214996

STUDY DESIGN:
Intervention Model Description: Part A: Phase I study - Dose-escalation of RMC-4630 and LY3214996 combination to determine RP2D/MTD.
  Dose level will be escalated according to standard 3+3 design.
  Part B: Phase Ib study - To further characterize the safety, tolerability and PK/PD of the RP2D of the RMC-4630 and LY3214996 combination.
  Expansion cohort in which patients with KRASm PDAC will be treated with the RP2D found in Part A of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase I - Dose-escalation (Experimental): This is a single-center open-label phase I dose-finding study (3+3 classical design) evaluating the RP2D of RMC-4630 in combination with LY3214996. Based on the safety, tolerability, and PK and PD data from the dose-finding stage of the study, a RP2D will be defined for the expansion phase.
  Interventions: Drug: RMC-4630; Drug: LY3214996
- Phase Ib (Experimental): The phase Ib expansion cohort study is intended to further characterize the safety, tolerability and PK/PD of the selected dose of RMC-4630 in combination with LY3214996 in patients with advanced KRASm PDAC. Furthermore, it will explore the clinical activity of RMC-4630 in combination with LY3214996 in patients with advanced KRASm PDAC.
  Interventions: Drug: RMC-4630; Drug: LY3214996

INTERVENTIONS:
Drug: RMC-4630 — * SHP2-inhibitor
  * Powder in capsule
  * Administered on day 1 and day 2 of every week
  Other Names: SAR442720
Drug: LY3214996 — * ERK inhibitor
  * Powder in capsule
  * Administered every day

SUMMARY:
This is a Phase I/Ib study in which the safety of the combination therapy of RMC-4630 and LY3214996 in the treatment of KRAS mutant cancers will be studied.

DETAILED DESCRIPTION:
This is a phase I / Ib study in which the safety of the combination therapy of RMC-4630 and LY3214996 in the treatment of KRAS mutant cancers colorectal cancer (CRC), non-small cell lung cancer (NSCLC) and pancreatic ductal adenocarcinoma will be studied.

The phase I dose-escalation study is designed to identify the recommended phase 2 dose (RP2D) of the combination regimen of RMC-4630 (SHP2-inhibitor) plus LY3214996 (ERK-inhibitor) in patients with KRASm CRC, NSCLC or PDAC.

The phase Ib expansion cohort is designed to further characterize the safety of the selected dose from the first stage of the study and to explore the clinical activity of RMC-4630 in combination with LY3214996 in patients with metastatic KRASm PDAC.

ELIGIBILITY:
Inclusion Criteria:

1. Part A: Histological or cytological proof of advanced KRASm NSCLC, CRC or PDAC; PART B: Histological or cytological proof of advanced KRASm PDAC.
2. Age => 18 years;
3. Able and willing to give written informed consent;
4. WHO performance status of 0 or 1
5. Able and willing to undergo blood sampling for PK and PD analysis;
6. Able and willing to undergo tumor biopsies prior to start (or have undergone a biopsy within 2 months of inclusion), while on study treatment and upon progression of disease;
7. Life expectancy => 3 months and no deterioration or hospitalizations within 2 weeks leading to C1D1, allowing adequate follow up of toxicity evaluation and antitumor activity;
8. Evaluable disease according to RECIST 1.1 criteria; (PART A and PART B);
9. Women of childbearing potential must have a negative serum pregnancy test within 14 days prior to registration and agree to use effective contraceptive methods, as defined in section 5.9.3, through-out the treatment period, and for 4 months after the study treatment
10. Adequate organ system function.

Exclusion Criteria:

1. Part A: No excluded genotypes

   Part B: Excluded genotypes (including co occurring mutations):
   * NRAS (except G12A/C)
   * RASQ61
   * KRASG13
   * BRAF Class 1, 2, or unclassified
   * PIK3CA
   * STK11
   * KEAP1
2. Any treatment with investigational drugs within 30 days prior to receiving the first dose of investigational treatment;
3. Patients currently using concomitant medication that are strong inhibitors or inducers of CYP3A4;
4. History of another malignancy Exception PART A: Patients who have been disease-free for at least 3 years, or patients with a history of completely resected non-melanoma skin cancer and/or patients with indolent completely resected second malignancies are eligible. Exception PART B: Adequately treated carcinoma in situ of the cervix and adequately treated basal cell carcinoma of the skin.
5. Symptomatic or untreated leptomeningeal disease
6. Symptomatic brain metastasis. Patients previously treated or untreated for these conditions that are asymptomatic in the absence of corticosteroid and anticonvulsant therapy (for at least 4 weeks) are allowed to enroll. Radiotherapy for brain metastasis must have been completed at least 6 weeks prior to start of study treatment. Brain metastasis must be stable with verification by imaging (e.g.

   brain MRI or CT completed at screening demonstrating no current evidence of progressive brain metastases). Patients are not permitted to receive antiepileptic drugs or corticosteroids.
7. Patients who have had previous treatment with any targeted drug combination known to interfere RAS/MEK/MAPK pathway components.
8. Toxicities related to prior treatments > grade 1 (excluding alopecia)
9. History of interstitial lung disease or pneumonitis
10. Woman who are breast feeding;
11. Patients who have undergone any major surgery within the last 4 weeks prior to starting study drug or who would not have fully recovered from previous surgery.
12. Radio- or chemotherapy within the last 4 weeks prior to receiving the first dose of investigational treatment; except a palliative dose of radiation of 8 Gy, which is allowed up to one week before study start and should not be applied to the target lesion.
13. Uncontrolled infectious disease or known Human Immunodeficiency Virus HIV-1 or HIV-2 type patients;
14. Patients with a known history of or uncontrolled hepatitis B (HBV) or C (HCV);
15. Patients with known alcoholism, drug addiction and/or psychiatric of physiological condition which in the opinion of the investigator would impair study compliance;
16. Patients with cardiac comorbidities (myocardial infarct within 6 months of study start, NYHA class ≥ III, congestive heart failure or instable angina pectoris), uncontrolled hypertension (systolic blood pressure > 160 mm Hg and/or diastolic pressure > 90 mm Hg), prolonged QT interval(> 440 ms for men, > 460 ms for women) or patients who have had a stroke within 6 months prior to start study.
17. Other severe, acute, or chronic medical or psychiatric condition, laboratory abnormality active infections that may increase the risk associated with study participation or study drug administration or that may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for the study.
18. Patients with pulmonary embolisms or deep venous thrombosis (DVT) within 3 months prior to start
19. Known hypersensitivity to one of the study drugs or excipients.
20. Baseline diarrhea and/or any condition that would impair absorption of oral agents
21. Patient with a history or findings of central or branch retinal artery or venous occlusion with significant vision loss or other retinal diseases that cause current visual impairment or would likely cause visual impairment over the time period of the study, as assessed by an ophthalmologist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Phase I - Maximum tolerated dose (MTD) | Through study completion, an average of 2 year
  Maximum Tolerated Dose (MTD) of the combination of RMC-4630 and LY3214996. Dose escalation will follow 3+3 design. The CTCAE criteria will be used to determine if adverse events and lab abnormalities will be accounted as dose limiting toxicity (DLT)
Phase Ib - Clinical activity of the RMC-4630 and LY3214996 combination in patients with KRASm PDAC | Tumor assessed every 8 weeks through study completion, with an expected average of 4 treatment cycles (each cycle is 28 days)
  Response and progression evaluated using internationally accepted response criteria and definitions proposed by the RECIST criteria

SECONDARY OUTCOMES:
Observed plasma concentrations of RMC-4630 and LY3214996 | Prior to initial dose on day 1, day 8, day 15, day 22 and 0.5, 1, 2, 4, 8, 24 hours post dose on day 1 and day 15.
  Blood samples are obtained and plasma concentrations of RMC-4630 and LY3214996 are measured using a validated LC-MS/MS method.
Area under de plasma - time concentration curve of RMC-4630 and LY3214996 | Prior to initial dose on day 1, day 15, and 0.5, 1, 2, 4, 8, 24 hours post dose.
  Blood samples are obtained and plasma concentrations of RMC-4630 and LY3214996 are measured using a validated LC-MS/MS method.
Elimination half-life of RMC-4630 and LY3214996 (T1/2) | Prior to initial dose on day 1, day 15, and 0.5, 1, 2, 4, 8, 24 hours post dose.
  Blood samples are obtained and plasma concentrations of RMC-4630 and LY3214996 are measured using a validated LC-MS/MS method.
Total body clearance of RMC-4630 and LY3214996 | Prior to initial dose on day 1, day 15, and 0.5, 1, 2, 4, 8, 24 hours post dose.
  Blood samples are obtained and plasma concentrations of RMC-4630 and LY3214996 are measured using a validated LC-MS/MS method.
Volume of distribution of RMC-4630 and LY3214996 | Prior to initial dose on day 1, day 15, and 0.5, 1, 2, 4, 8, 24 hours post dose.
  Blood samples are obtained and plasma concentrations of RMC-4630 and LY3214996 are measured using a validated LC-MS/MS method.
Baseline molecular status of potential predictive markers of tumor response | Before start of treatment, during treatment and (optional) after treatment discontinuation with RMC-4630 and LY3214996 with an expected average of 4 treatment cycles (each cycle is 28 days)
  Baseline molecular status of potential predictive markers of tumor response wil be studied in tumor biopsies taken before treatment, during treatment and (optional) after treatment using the Ampliseq SOCV1panel
Pharmacodynamic biomarkers of RMC-4630 and LY3214996 | Before start of treatment, during treatment and (optional) after treatment discontinuation with RMC-4630 and LY3214996 with an expected average of 4 treatment cycles (each cycle is 28 days)
  To evaluate pharmacodynamic (PD) biomarkers of the RMC-4630- LY3214996 combination, the expression levels of relevant down-stream proteins are measured in tumor biopsies, using the Ampliseq SOCV1panel. Markers to be assessed include molecular status (mutation/amplification/expression) of markers related to the RAF/MEK/ERK and PI3K/AKT pathway (e.g. BRAF, HRAS, NRAS, KRAS, PIK3CA, PTEN, pS6-RP, c-MET, EGFR, HER-3, pERK, pAKT, pEGFR, and pRSK).
Potential mechanism of resistance | Before start of treatment, during treatment and (optional) after treatment discontinuation with RMC-4630 and LY3214996 with an expected average of 4 treatment cycles (each cycle is 28 days)
  Potential mechanisms of are studied in tumor biopsies taken before treatment, during treatment and (optional) after treatment using the Ampliseq SOCV1panel

CONTACTS AND LOCATIONS:
Overall Officials: Emile Voest, MD, PhD, Study Director — Netherlands Cancer Institute - Antoni van Leeuwenhoek
Locations (1):
- Netherlands Cancer Institute - Antoni van Leeuwenhoek, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mainardi S, Mulero-Sanchez A, Prahallad A, Germano G, Bosma A, Krimpenfort P, Lieftink C, Steinberg JD, de Wit N, Goncalves-Ribeiro S, Nadal E, Bardelli A, Villanueva A, Bernards R. SHP2 is required for growth of KRAS-mutant non-small-cell lung cancer in vivo. Nat Med. 2018 Jul;24(7):961-967. doi: 10.1038/s41591-018-0023-9. Epub 2018 May 28. PMID 29808006
- [Derived] Frank KJ, Mulero-Sanchez A, Berninger A, Ruiz-Canas L, Bosma A, Gorgulu K, Wu N, Diakopoulos KN, Kaya-Aksoy E, Ruess DA, Kabacaoglu D, Schmidt F, Kohlmann L, van Tellingen O, Thijssen B, van de Ven M, Proost N, Kossatz S, Weber WA, Sainz B Jr, Bernards R, Algul H, Lesina M, Mainardi S. Extensive preclinical validation of combined RMC-4550 and LY3214996 supports clinical investigation for KRAS mutant pancreatic cancer. Cell Rep Med. 2022 Nov 15;3(11):100815. doi: 10.1016/j.xcrm.2022.100815. PMID 36384095